CLINICAL TRIAL: NCT05791734
Title: Validation of Preoperative Shower Quality Assessment by ATPmetry
Brief Title: Validation of Preoperative Shower Quality Assessment by ATPmetry (PRODOUCH'Eval)
Acronym: PRODOUCH'Eval
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/0178/OB
Record Dates: First submitted 2023-02-28; First posted 2023-03-30 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Ambulatory Surgical Procedures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- assessing preoperative skin cleanliness: 2 skin swabs for ATPmetry measurement and direct skin visual observation by a nurse
  Interventions: Other: assessing preoperative skin cleanliness

INTERVENTIONS:
Other: assessing preoperative skin cleanliness — 2 skin swabs on surgical incision sites and direct skin visual observation by a nurse

SUMMARY:
According to the 2013 guidelines of the French Society for Hospital Hygiene (SF2H), it is recommended to carry out at least one preoperative shower, with an antiseptic soap or a mild soap as close as possible to the operation. This preoperative shower aims to eliminate dirt and make the skin clean to facilitate the subsequent action of the antiseptic in the operating theatre. Thus, detersion is no longer carried out systematically but is only recommended in the presence of soiled skin. The preoperative shower, and the verification of its effectiveness, therefore become essential steps in the preoperative skin preparation. Indeed, the cleanliness of the skin influences the quality of the antisepsis performed in the operating theatre.

Visual assessment of preoperative skin cleanliness by the nurse is currently the reference technique. However, a qualitative pilot study (Consiglio et al., Rech Soins Inf 2021) of nine obese patients and eleven surgical nurses revealed a lack of visual verification of skin cleanliness, which caregivers found difficult to perform. In a second multicentre study of 430 patients (Boulet et al., under review by Nursing Open), only 17% reported visual verification of skin cleanliness. Thus, this initial work highlights a barrier for caregivers to visually check preoperative skin cleanliness.

The ATPmetry method was initially developed to assess the cleanliness of surfaces. In a second phase, the manufacturer (Hygiena®) showed through a study of 20 professionals that this method also allowed the evaluation of skin cleanliness of hands after washing. This method would have the advantage of being objective, potentially improving acceptability to caregivers and patients compared to direct visual inspection of skin cleanliness. Thus, ATPmetry appears to us as a method of interest for assessing preoperative skin cleanliness, but needs to be validated for this indication.

To date, there is no other method than the simple subjective visual skin assessment by the caregiver, which is highly exposed to a bias of non-reproducibility and inter-observer variability.

DETAILED DESCRIPTION:
This study aims to evaluate a simple and objective method of measuring preoperative skin cleanliness (by swabbing and ATPmetry), in order to eventually standardise this method for routine practice.

The reproducibility of the ATPmetry measurement will be assessed as well as its concordance with two other methods (visual skin inspection and visual swab inspection). An statistical analysis will assess its agreement with each of the other two methods, as compared to the agreement between the two methods.

ELIGIBILITY:
Inclusion Criteria:

Patients inclusion criteria:

* Age greater than or equal to 18 years
* patient with ambulatory surgical procedures
* Patient scheduled for a surgical procedure for which the incision site is cutaneous
* Patient covered by national health insurance
* Patient having read and understood the information letter and having expressed oral non-opposition to the research

Exclusion Criteria:

The following patients will be excluded from the study

* Patients scheduled for a surgical procedure with a muqueous incision site
* patients < 18 ans
* Pregnant or breastfeeding women
* Patients who have not given their consent to participate or are unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with ambulatory surgical procedures
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
innovative method | before surgery
  preoperative skin cleanliness as assessed by ATPmetry
reference method | before surgery
  preoperative skin cleanliness as assessed by direct visual observation by a nurse

SECONDARY OUTCOMES:
visual observation | before surgery
  Visual observation of the cleanliness of one of the two swabs before analysis by ATPmetry. This immediate observation will be made by a second nurse (unaware of the first nurse's judgement of skin cleanliness), who will assess skin cleanliness as "unsatisfactory" if the swab is stained.

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No